CLINICAL TRIAL: NCT06135753
Title: Psychosomatic Assessment and Intervention in Fibromyalgia
Brief Title: Psychosomatic Intervention in Fibromyalgia.
Acronym: PSY-FM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Fiammetta Cosci, Associate Professor in Clinical Psychology, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY-FM
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Psychosomatic Intervention; Cognitive Restructuring; Museum Therapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: This is a pilot study, designed as a cross-sectional observation study (study 1) and as a randomized (1:1) controlled trial, comparing a multidisciplinary psychosomatic intervention based on cognitive restructuring vs a control condition both followed by museum therapy (study 2). The participants will receive a baseline psychosomatic assessment to confirm the diagnosis of fibromyalgia, then socio-demographic information, information on pharmacological/non-pharmacological treatments, on the history of medical diseases and on the psychological status will be collected. Thereafter, the subjects will be randomly assigned to experimental group or to a control condition. The subjects will be re-assessed at the end of session 4, and at the end of session 7, 8, 9 of museum therapy and at 3 and 6-month follow-up.
Who Masked: Participant
Masking Description: Participants will not be informed if they will receive the psychosomatic intervention or the control condition. At the end of the study they will receive this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: psychosomatic intervention based on cognitive restructuring followed by Museum Therapy (Experimental): A psychosomatic intervention based on cognitive restructuring will be used as the non-pharmacological therapeutic strategy and 4 sessions will be delivered every other week with a duration of 120 minutes each in a group format with 10 participants.
  The museum therapy will include 4 sessions, directed by the clinical psychologist and a museum educator, aimed at facilitating emotional expressions and participants' behavioral activation. The sessions will be delivered starting 2 weeks after the last session of the psychosomatic intervention as part of the Benessere al Museo Project by Uffizi Galleries.
  A final additional session will be proposed.
  Interventions: Other: psychosomatic intervention based on cognitive restructuring.; Other: Experimental and control condition: Museum therapy
- Placebo Comparator: Control condition followed by Museum Therapy (Placebo Comparator): The control condition will include 4 every other week sessions based on Lifestyle and well-being National Institute for health and Care Excellence (NICE) Guidelines (https://www.nice.org.uk/guidance/lifestyleandwellbeing) and on World Health Organization 12 steps to healthy eating (http://www.euro.who.int/en/health-topics/disease-prevention/nutrition/a-healthylifestyle). These sessions will inform participants about well-being and lifestyles which can influence it.
  The museum therapy will include 4 sessions, directed by the clinical psychologist and a museum educator, aimed at facilitating emotional expressions and participants' behavioral activation. The sessions will be delivered starting 2 weeks after the last control group's session as part of the Benessere al Museo Project by Uffizi Galleries.
  A final additional session will be proposed.
  Interventions: Behavioral: Control condition; Other: Experimental and control condition: Museum therapy

INTERVENTIONS:
Other: psychosomatic intervention based on cognitive restructuring. — Participants will receive information on psychosomatic phenomena and over-listening of somatic manifestations (Session 1), interpretation and possible catastrophization of somatic manifestations even when they might be well-known health problems or potential physiological or para-physiological manifestations (Session 2), pain-proneness (Session 3) and mental pain and psychological distress in somatizers (Session 4). The second part of each session will be devoted to group cognitive restructuring, thus participants will be stimulated in verifying how the phenomena illustrated are in their lives and how they can be differently conceptualized in order to be less intrusive and less able to reduce their own functioning.
  Arms: Experimental: psychosomatic intervention based on cognitive restructuring followed by Museum Therapy
Behavioral: Control condition — The control condition will include 4 sessions that will inform participants about well-being and lifestyles which can influence it. They will be articulated as follows. Session 1: illustrating the concept of lifestyle and well-being. Session 2 and session 3: illustrating healthy eating and steps to healthy eating. Session 4: illustrating physical exercise and how it promotes health.
  Arms: Placebo Comparator: Control condition followed by Museum Therapy
Other: Experimental and control condition: Museum therapy — Session 5-6-7: preselected painting works from the Uffizi Galleries (Florence) will be presented to the participants in order to trigger reflections and emotional responses on specific pain related topics. Session 8: visit the Galleria di Arte Moderna at Palazzo Pitti, in person. Each session will be aimed at facilitating emotional expressions and partecipants' behavioral activation and identifying thoughts associated with those emotions and, if appropriate, remodulating them in a functional way (cognitive restructuring).
  Session 9: share the experience of the previous meetings and to recap strategies and skills which could be implemented in FM participants' daily life to cope with their illness.

SUMMARY:
Fibromyalgia is a widespread musculoskeletal pain syndrome. It is characterized by physical manifestations which are also the expression of a psychological distress as well as specific illness attitudes and behaviors. Indeed, it is considered a psychosomatic disorder. In this framework, we hypothesize the clinical utility of a psychosomatic assessment guided by rheumatologists and clinical psychologists (Study 1) and the utility of an integrated multidisciplinary psychosomatic intervention based on cognitive restructuring/psychoeducation followed by museum therapy (Study 2). For Study 1 a cross-sectional observation study will be implemented, for Study 2 a randomized controlled trial will be applied.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a widespread musculoskeletal pain syndrome characterized by chronic widespread pain, unrefreshing sleep, physical exhaustion, and cognitive difficulties. It occurs in all populations throughout the world, with prevalence between 2% and 4% in general populations. Definition, pathogenesis, diagnosis, and treatment of FM remain points of contention. There is no specific diagnostic laboratory test or biomarker to support the diagnostic process and the diagnosis is clinical. For this reason, rheumatologists and clinical psychologists are strongly involved in the diagnostic process and might benefit from tools for comprehensive psychosomatic assessment. Also the treatment of FM remains a challenge, because pharmacological interventions don't consider psychological and social problems and non-pharmacological treatments have shown poor efficacy and are often tested via non-rigorous methods. A multidisciplinary approach which include biological aspects and psychological one, under comprehensive psychosomatic principles, seem to be the best choice for FM.

The primary aim of the present study is to evaluate the psychological status of FM subjects, focusing on a psychosomatic assessment and then testing the efficacy of a multidisciplinary psychosomatic intervention based on cognitive restructuring followed by museum therapy vs a control condition followed by museum therapy.

ELIGIBILITY:
Inclusion Criteria:

1. able and interested in participating to the research, as proved by signed Informed consent;
2. a diagnosis of FM according to the Italian Society for Rheumatology clinical practice guidelines (Ariani et al., 2021)
3. age higher than 18 years

Exclusion Criteria:

1. co-occurrence of psychiatric disorder(s) according to the Diagnostic and Statistical Manual of mental disorders, 5th edition (American Psychiatric Association, 2013) as diagnosed via the Mini-International Neuropsychiatric Interview;
2. currently under psychotherapy;
3. pharmacological modifications during the period of the trial;
4. undergoing non pharmacological interventions during the period of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Psychosomatic status | change from baseline to 9-session of treatment
  Diagnostic Criteria for Psychosomatic Research-Revised Semi-Structured Interview (Fava et al., 2017)
Level of distress, well-being and quality of life | change from baseline to 6-month follow up
  The PsychoSocial Index (Piolanti et al., 2016)

SECONDARY OUTCOMES:
Psychiatric status | change from baseline to 9-session of treatment
  Mini-International Neuropsychiatric Interview (Sheehan et al., 1998)
Psychological distress | change from baseline to 6-month follow up
  Symptom Questionnaire (Fava et al., 1983); (min: 0, max: 92, the highest score corresponds to the highest level of psychological distress)
Mental pain | change from baseline to 6-month follow up
  Mental Pain Questionnaire (Fava, 2016); (min: 0, max: 20, the highest score corresponds to the highest level of mental pain)
Feelings of loneliness and social isolation | change from baseline to 6-month follow up
  the UCLA Loneliness Scale (Russell et al., 1980); (20 items, the highest score corresponds to the highest level of feelings of lolliness)
Well-being | change from baseline to 6-month follow up
  World Health Organization-Five Well-Being Index (min: 0, max: 25, the highest score corresponds to the lowest level of well-being)

CONTACTS AND LOCATIONS:
Overall Officials: Fiammetta Cosci, MD, Prof.ssa, Principal Investigator — University of Florence
Locations (1):
- Rheumtoi Unit, Academic Hospital Careggi, Florence, Italia/firenze, Italy

IPD SHARING:
Plan to Share IPD: No